CLINICAL TRIAL: NCT02468492
Title: Synovial Fluid Biomarker and Mesenchymal Stem Cell Response to PRP in Knee Osteoarthritis With Clinical and Imaging Outcome Correlation: Proof of Concept Study
Brief Title: Pilot Synovial Fluid Molecular/Stem Cell Response to PRP in Knee Osteoarthritis: Clinical & Imaging Outcome Correlation
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Hunter Holmes Mcguire Veteran Affairs Medical Center (U.S. Federal Agency)
Collaborators: Foundation for Physical Medicine and Rehabilitation (Other)
Responsible Party: Principal Investigator, Dr. Lance Goetz, Staff Physician, Hunter Holmes Mcguire Veteran Affairs Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB #01979/FDA IDE#15944
Record Dates: First submitted 2015-05-31; First posted 2015-06-10 (Estimated); Last update posted 2017-08-16 (Actual); Status verified 2017-08

CONDITIONS: Knee Osteoarthritis
Keywords: Knee Osteoarthritis; Platelet Rich Plasma; Mechanism of Action; Stem Cells; Synovial Fluid
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Platelet Rich Plasma (Experimental): Approximately 5mL of intraarticular PRP once at baseline
  Interventions: Biological: Platelet Rich Plasma
- Normal Saline (Other): Approximately 5mL of intraarticular normal saline once at baseline
  Interventions: Other: Normal Saline

INTERVENTIONS:
Biological: Platelet Rich Plasma — Platelet rich plasma injection into knee versus placebo (saline) injection.
  Other Names: Platelet Concentrate
  Arms: Platelet Rich Plasma
Other: Normal Saline — Platelet rich plasma injection into knee versus placebo (saline) injection.
  Arms: Normal Saline

SUMMARY:
The purpose of this study is to evaluate the affect that platelet rich plasma has on the molecular an cellular functioning of the knee joint.

DETAILED DESCRIPTION:
In this study 18 subjects with mild to moderate symptomatic knee osteoarthritis will be recruited per an IRB approved protocol with explicit inclusion and exclusion criteria. Subjects who are enrolled and meet all criteria will be blinded and randomized (2:1) to receive Platelet Rich Plasma or normal saline "control". Prior to the intervention, a synovial fluid aspiration will occur. At follow up number one (approximately 10 days from baseline) a repeat aspiration will occur and a differential analysis of the molecular and biochemical effects will be undertaken; this data will serve as the primary outcome measures. This data will be correlated to clinical and imaging outcome measures which will be secondary outcome measures completed at baseline and intermittently throughout the study. The duration of the study is one year.

ELIGIBILITY:
Inclusion Criteria:

1. Early/Mild to Moderate Stage knee osteoarthritis (KOA), as determined by Kellgren-Lawrence Grade 2 to 3 on PA standing radiograph within the past three months;

   * A prospective subject who has a diagnosis of non-end stage KOA (i.e., a potential study candidate) and expresses interest in participating but has no XRAY within the specified time-period will be sent for a fresh XRAY. This XRAY will be read by a radiologist & be paid for by the study.
2. >=40 years of age;
3. Average 100-point VAS score of >50, on average, within the past 3 months*, with KOA felt to be the primary contributor to pain.

   * Alternate 10-point scales with pain scores averaging >5 may be considered if the prospective subject also completes a VAS with score >50 at screening.
4. Exam consistent with KOA being primary etiology of pain;
5. No signs of inflammatory arthropathy in medical record, history or physical examination;
6. A >3 millimeter intra-articular (IA) effusion present on ultrasound evaluation.
7. [If a chronic liver or renal disease patient, evidence of stable disease over/within the past six months, else exclusion.]
8. Veteran receiving care at McGuire VAMC.

Exclusion Criteria:

1. Morbid obesity (BMI >40);
2. Poorly controlled diabetes (hemoglobin A1C > 7.5 or fasting blood glucose of >200) in last 6 months;
3. Ipsilateral knee surgery, trauma within last 6 months, or corticosteroid injection within 3 months.
4. 4. History of inflammatory arthropathy (RA, SLE or crystalline arthritis of the knee)**;
5. Any rheumatoid arthritis or gout diagnosis is exclusionary.
6. Current infection of the affected joint or any other uncontrolled or untreated active infection.
7. Moderate to severe anemia (hemoglobin < 11 g/dl) or thrombocytopenia (platelet count < 100,000); Hemoglobin >17 g/dl or <11 g/dl and/or platelet counts >500,000 or <100,000 platelets/μl.

   * [CBC obtained within 6 months will be required, even if obtained at initial screening visit.]
8. Individuals on dialysis, with liver failure, or uncontrolled renal or liver disease are excluded.

   * In those with chronic renal or liver disease, documentation of stable disease within the most recent 6 months will be required.
9. Individuals on a therapeutic anticoagulant (e.g., Warfarin, Dabigatran, Enoxaparin) and those with a history of coagulopathy are excluded.

   * Per standard clinical practice, subjects on anti-platelet therapy are not excluded.
10. Pregnancy or breast-feeding;

    * Female subjects of child-bearing potential must have a negative pregnancy screen prior to enrollment.
    * Female subjects of child-bearing potential must confirm they are not actively breast-feeding prior to enrollment.
11. Current illicit drug abuse / active alcohol abuse (i.e, Current substance abuse);
12. Uncontrolled psychiatric disorder;
13. Lack of transportation (i.e., to get to/from appointments at VAMC) and/or willingness to attend study appointments (screening/consent, Intervention, Day10-follow-up, Month-6 follow-up, and then visits over-the-phone / in-person / or via Telehealth for Month-3 and Month-12;
14. Advanced or currently active cancer.
15. Blood disorders (such as Sickle Cell Anemia, TTP, others)
16. Vulnerable populations: Individuals incapable of making informed decisions will not be enrolled, nor will those under some form of incarceration.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-09; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Biochemical Molecular Outcomes | Baseline and 10 day follow up
  Evaluate for change in biochemical molecular milieu temporal response after PRP injection or normal saline (control) compared to baseline, as measured by multiplex suspension array technology.

SECONDARY OUTCOMES:
Clinical Outcomes | 1 year
  Evaluation for change in pain level via VAS and WOMAC at baseline and follow up.
Imaging Outcomes | 6 months
  Evaluation for change in joint space width using knee radiographs at baseline and 6 month follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Lance L Goetz, MD, Principal Investigator — Hunter Holmes McGuire VAMC
Locations (1):
- Hunter Holmes McGuire VA Medical Center, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided
Publications planned.